CLINICAL TRIAL: NCT06120127
Title: Postoperative Chemotherapy With/Without Radiotherapy and Immunotherapy for Colorectal Liver Metastases With High Risk of Locally Recurrence: A Randomized Controlled Phase II Trial
Brief Title: Postoperative Chemotherapy With/Without Radiotherapy and Immunotherapy for Colorectal Liver Metastases With High Risk of Locally Recurrence
Acronym: IMPROVE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2023-258-3377
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Radiotherapy; Immunotherapy; Liver Metastases; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiotherapy; Drug Therapy; spartalizumab; sintilimab

STUDY DESIGN:
Intervention Model Description: adjuvant radiotherapy: SBRT; immunotherapy: sintilimab chemotherapy: XELOX
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chemotherapy with radiotherapy and immunotherapy (Experimental): radiotherapy: SBRT of liver lesions; postoperative chemotherapy and immunotherapy: chemotherapy by investigators' choice with sintilimab for 18 weeks
  Interventions: Radiation: SBRT; Drug: Chemotherapy; Drug: PD-1 antibody
- chemotherapy (Active Comparator): postoperative chemotherapy: chemotherapy by investigators' choice for 18 weeks
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Radiation: SBRT — postoperative SBRT of liver lesions
  Other Names: radiotherapy
  Arms: chemotherapy with radiotherapy and immunotherapy
Drug: Chemotherapy — XELOX/FOLFOX/FOLFIRI
Drug: PD-1 antibody — Sintilimab (200mg d1，q3w)
  Other Names: Sintilimab
  Arms: chemotherapy with radiotherapy and immunotherapy

SUMMARY:
This study is a randomized controlled phase II trial to evaluate the efficacy of the combination of stereotactic body radiation therapy (SBRT) and immunotherapy with postoperative chemotherapy in colorectal cancer liver metastasis (CRLM) patients with high risk of locally recurrence. Researchers will compare the combination therapy with the postoperative chemotherapy alone to see if postoperative chemotherapy plus SBRT and immunotherapy can further reduce the risk of recurrence and metastasis after surgery.

DETAILED DESCRIPTION:
40-50% of colorectal cancer patients have metastases at the time of diagnosis, of which liver metastases are the most common. Surgical resection is the most likely cure for CRLM patients, however, more than 50% of patients will experience recurrence within 2 years after resection of liver metastases. SBRT can be an effective and safe treatment modality, which can not only provide better local control of metastatic lesions, but also has a sensitizing immunotherapeutic effect. SBRT can effectively synergize with anti-PD-1/PD-L1 antibodies to activate the immune microenvironment of CRLM patients and improve survival. However, in CRLM patients after surgery, whether combining SBRT, immunotherapy and adjuvant chemotherapy results in better survival than chemotherapy alone, the evidence is insufficient.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years old, female and male
2. pathological and imaging confirmed colorectal colorectal liver metastases (synchronous or heterochronous)
3. Metastatic liver lesions <= 5
4. Primary colorectal cancer under control
5. Absence of evidence of extra-hepatic diseases
6. Metastatic liver lesions received resection with insufficient margin (<0.5cm) or R1/R2 resection
7. Karnofsky >= 70
8. Adequate organ function without contraindications to surgery, radiotherapy and immunotherapy
9. Without previous antitumoral immunotherapy
10. With good compliance
11. Signed the inform consent

Exclusion Criteria:

1. Pregnancy or breast-feeding women
2. History of other malignancies within 5 years (except cured skin cancer and cervical cancer in situ)
3. History of uncontrolled epilepsy, central nervous system disease, or psychiatric disorders
4. Clinically serious heart disease, such as symptomatic coronary artery disease, New York Heart Association (NYHA) class II or worse congestive heart failure or severe arrhythmia requiring pharmacologic intervention, or history of myocardial infarction within the last 12 months
5. Immunodeficiency disease, autoimmune diseases or long-term using of immunosuppressive agents
6. Severe uncontrolled recurrent infections
7. Baseline blood and biochemical indicator do not meet the following criteria: neutrophils >=1.5×10^9/L, Hb >=90g/L, PLT >=100×10^9/L, ALT/AST<=2.5 ULN, Cr <= 1ULN
8. Allergic to any component of the therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From the date of randomization until the date of first documented progression or date of death from any cause, whichever come first, assessed up to 12 months
  Evaluate the effect of the combination of adjuvant chemotherapy, SBRT and immunotherapy versus observation on progression free survival

SECONDARY OUTCOMES:
Local control rate | From the date of randomization until the date of first documented locally tumor recurrence, assessed up to 12 months
  To evaluate local control rate after the combination of adjuvant chemotherapy, SBRT and immunotherapy in comparison to observation alone
Overall survival | From date of randomization until the date of death from any cause, assessed up to 36 months
  To evaluate overall survival after the combination of adjuvant chemotherapy, SBRT and immunotherapy in comparison to observation alone
Grade 3-4 adverse effect rate | From date of randomization until the date of death from any cause, assessed up to 3 years
  Rate of chemotherapy, SBRT and immunotherapy related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Fan Xia, M.D,PH.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China